CLINICAL TRIAL: NCT02368301
Title: An Expanded Access Program for Elotuzumab in Combination With Lenalidomide Plus Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Expanded Access Treatment Protocol CA204-143
Status: No longer available | Type: Expanded Access
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA204-143
Record Dates: First submitted 2015-02-06; First posted 2015-02-23 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — elotuzumab; Lenalidomide; Dexamethasone

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Elotuzumab in combination with Lenalidomide and Dexamethasone — Elotuzumab in Combination With Lenalidomide Plus Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma

SUMMARY:
The objective of this expanded access program is to provide treatment with elotuzumab in combination with lenalidomide and dexamethasone for patients with relapsed or refractory multiple myeloma at U.S. sites where licensed physicians determine clinical need.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria

* Men and women 18 years and older.
* Active, relapsed or refractory multiple myeloma by IMWG (International myeloma Working Group) criteria as assessed by the treating physician and have received one prior line of multiple myeloma therapy.
* Prior lenalidomide exposure is permitted only if they fulfill all of the following:.

  i) Were not refractory to prior lenalidomide defined as no progression while receiving lenalidomide (induction dose) or within 60 days of last dose of lenalidomide. Patients progressing on lenalidomide maintenance dose are eligible for enrolment.

A. Patient did not discontinue lenalidomide due to a Grade ≥ 3 related AE.

Exclusion Criteria

* Active plasma cell leukemia (defined as either 20% of peripheral WBC comprised of plasma/CD138+ cells or an absolute count of 2 x 109/L).
* All Adverse Events of any prior chemotherapy, surgery, or radiotherapy not resolved to NCI CTCAE (v. 3.0) Grade ≤ 2.
* Significant cardiac disease as determined by the treating physician including cardiac amyloidosis.
* HIV infection or active hepatitis A, B, or C.
* History of participation in elotuzumab studies CA204-004, CA204-006 or CA204-009.
* Inadequate recovery from prior surgery or prior myeloma therapy. If prior allogeneic stem cell transplant, history of moderate to severe chronic graft versus host disease (GvHD).
* Any medical conditions that, in the attending physician's opinion, would impose excessive risk to the patient.
* Certain abnormal physical or laboratory findings.
* Hypersensitivity to lenalidomide, dexamethasone, any excipients in the elotuzumab formulation, or recombinant protein.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: EAP Investigator Requests — http://www.bms.com/clinical_trials/investigator_sponsored_research/Pages/expanded-access-program.aspx
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm